CLINICAL TRIAL: NCT06092879
Title: Scemblix® (Asciminib): Prospective Non Interventional Study as 3rd Line Therapy or More to Treat Adult Patients With CML-CP in Real World Setting in France
Brief Title: Asciminib Prospective Non Interventional Study as 3rd Line Therapy or More to Treat Adult Patients With CML- CP in Real World Setting in France
Acronym: ASSURE-3
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001AFR04
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; CML; asciminib; France
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Asciminib: Adult patients with Ph+ CML-CP previously treated with two or more tyrosine kinase inhibitors
  Interventions: Other: Asciminib

INTERVENTIONS:
Other: Asciminib — There is no treatment allocation. Patients administered Asciminib by prescription will be enrolled
  Other Names: Scemblix

SUMMARY:
The purpose of this study is to enhance the knowledge on asciminib treatment in a broader and real-life population by collecting additional data to characterize the treatment patterns of patients treated with asciminib, with a primary objective represented by maintenance on treatment at 12 months.

DETAILED DESCRIPTION:
The ASSURE-3 study is a national, multicentric, non-interventional, prospective study in real-life conditions with primary data collection in adult patients with Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase (Ph+ CML-CP) previously treated with two or more Tyrosine Kinase Inhibitors (TKIs). It will be conducted in France with hematologists, onco-hematologists, physicians with documented involvement in managing Ph+ CML-CP patients in routine practice, practicing in public or private health care institutions. Each patient will be followed during 15 months at M0, M1 and then every 3 months (rhythm of visits according to the routine clinical care), or until premature discontinuation of asciminib treatment.

Historical data will be abstracted retrospectively by the participating physicians from patient files, to collect information using an electronic case report form (eCRF). Primary data will be collected during inclusion and follow-up visits

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years at inclusion,
2. Patient with Ph+ CML-CP previously treated with two or more TKIs,
3. Patient for whom a decision has been taken by the treating physician (investigator) to initiate treatment with asciminib according to his own practice, the drug label / Summary of Product Characteristics (SmPC), and regardless of study participation,
4. Patient having given their non objection to participate to the study

Exclusion Criteria:

1. Patient with CML in accelerated phase (AP) or blastic phase (BP) at enrolment,
2. Patient with known history of T315I mutation,
3. Patient who previously received asciminib treatment,
4. Patient currently participating to an interventional clinical trial,
5. Patient with known contra-indication to asciminib according to the SmPC.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase (Ph+ CML-CP) previously treated with two or more tyrosine kinase inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients remaining on asciminib at 12 months | Month 12
  Proportion of patients remaining on asciminib treatment at 12 months to be provided

SECONDARY OUTCOMES:
Proportion of patients in major molecular response (MMR) - for patients not in MMR at treatment initiation | 12 months
  Molecular response to treatment: Response to treatment (MMR, BCR::ABL1 ≤ 0.1% on the International Scale, IS) at 12 months (+/- 1 month) for patients not in MMR at treatment initiation
Proportion of patients in MMR - for patients in MMR at treatment initiation | 12 months
  Molecular response to treatment: Maintenance of molecular response (MMR, BCR::ABL1 ≤ 0.1% on the International Scale, IS) at 12 months (+/- 1 month) for patients in MMR at treatment initiation
Proportion of patients in MR2, MMR, MR4.0, MR4.5, uMR4.5 - for all patients | 3 months, 6 months, 9 months, 12 months and 15 months
  Molecular response to treatment: Kinetics of response: MR2, MMR, MR4.0, MR4.5, undetectable MR4.5 for all patients.
  MR2, MR4, MR4.5 are defined as the transcript ratio of BCR-ABL1/ABL1 being 1% or less, 0.01% or less and 0.0032% or less respectively
BCR::ABL1 on the International Scale (IS) kinetics along treatment - for all patients | 15 months
  Kinetics of response: BCR::ABL1 on the International Scale (IS) for all patients
Time to MMR from the index date - for patients not in MMR at treatment initiation | Up to 15 months
  Kinetics of response: Time to MMR for patients not in MMR at treatment initiation
Time from the first MMR to the first loss of MMR - for patients not in MMR at treatment initiation | Up to 15 months
  Molecular response to treatment: Duration of MMR for patients not in MMR at treatment initiation
Event-Free Surviva (EFS) | Up to 15 months
  EFS: time from index date to occurrence of one the events listed among variables:
  * lack of efficacy, i.e., BRC::ABL1>1% or loss of CCyR if assessed
  * disease progression (CML-AP/BP, CML death)
  * death from any cause
  * definitive treatment discontinuation due to any reason
Progression-Free Survival (PFS) | Up to 15 months
  PFS: time from index date to occurrence of one of the progression markers listed among variables:
  * disease progression (CML-AP/BP, CML death),
  * death from any cause,
  * definitive treatment discontinuation due to any reason
Comorbidity profile | Baseline
  Charlson comorbidity index (CCI) at index date
Disease characteristics | Baseline
  Disease characteristics to be provided
History of TKI treatment | Baseline
  History of TKI treatment to be provided
Management of patients in real-life | 15 months
  Concomitant medications
Exposure patterns to asciminib | 15 months
  Exposure patterns to be provided
EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30) | Baseline, 3months, 6months, 9months, 12months, 15months
  The EORTC QLQ-C30 contains 30 questions assessed by the participant. There are 9 multiple-item scales: 5 scales that assess aspects of functioning (physical, role functioning, cognitive, emotional, and social); 3 symptom scales (Fatigue, Pain, and Nausea and Vomiting); and a global health status/Quality of Life (QOL) scale. There are 5 single-item measures assessing additional symptoms (i.e., dyspnea, loss of appetite, insomnia, constipation, and diarrhea) and a single item concerning perceived financial impact of the disease. All but two questions have 4-point scales ranging from "Not at all" to "Very much." The two questions concerning global health status/ QOL have 7 point scales with ratings ranging from "Very poor" to "Excellent." For each of the 14 domains, final scores are transformed such that they range from 0-100, where higher scores indicate improvement.
EORTC QLQ-CML24 questionnaire | Baseline, 3months, 6months, 9months, 12months, 15months
  The EORTC QLQ-CML24 was designed to supplement the QLQ-C30 - the QLQ-CML24 is not a stand-alone instrument but is to be used in conjunction with the QLQ-C30.
  The EORTC QLQ-CML 24 is composed of four multi-item scales and two single-item scales. The module consists of 24 items assessing symptoms burden (13 items), impact on worry/mood (4 items), impact on daily life (3 items), satisfaction with care and information (2 items) body image problems (1 item) and satisfaction with social life (1 item). The items were measured on four levels: 1=not at all, 2=a little, 3=quite a bit, 4=very much. For each domain, scores were averaged and transformed to 0 to 100. A higher score in satisfaction with social life domain indicates a higher level of satisfaction. A positive change from baseline indicates increasing satisfaction.
Emergence of mutations | Up to 15 months
  If available at end of treatment: mutational analysis, methods and results
Proportion of patient with an AE described during asciminib treatment among patient reporting the same AE which led to discontinuation with previous TKI treatments | Up to 15 months
  Cross intolerance with previous TKI treatments

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- France (55):
  - Novartis Investigative Site, Angers, France
  - Novartis Investigative Site, Challes-les-Eaux, France
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Saint Priest Jarez, Pays de la Loire Region
  - Novartis Investigative Site, Aix-en-Provence
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Antibes
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Brive-la-Gaillarde
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Cagnes-sur-Mer
  - Novartis Investigative Site, Cannes
  - Novartis Investigative Site, Castelnau-le-Lez
  - Novartis Investigative Site, Cesson-Sévigné
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Dunkirk
  - Novartis Investigative Site, Essey-lès-Nancy
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lens
  - Novartis Investigative Site, Libourne
  - Novartis Investigative Site, Lorient
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nevers
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Perpignan
  - Novartis Investigative Site, Périgueux
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Quimper
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Roubaix
  - Novartis Investigative Site, St-Malo
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Tarbes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Trévenans
  - Novartis Investigative Site, Troyes
  - Novartis Investigative Site, Valence
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Vesoul

IPD SHARING:
Plan to Share IPD: No